CLINICAL TRIAL: NCT04570345
Title: 3 Months Versus 12 Months Dual Antiplatelet Therapy After Second Generation Sirolimus Stent Implantation in ST-elevation Myocardial Infarction(BULK-STEMI)
Brief Title: 3 Months Versus 12 Months Dual Antiplatelet Therapy After Drug-eluting Stent Implantation in STEMI
Acronym: BULK-STEMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Kyungil Park, Associate professor, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAUHIRB-20-162
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Aspirin; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticagrelor monotherapy (Experimental): Ticagrelor monotherapy after 3-month DAPT(aspirin with ticagrelor)
  Interventions: Drug: ticagrelor monotherapy
- Aspirin with P2Y12 receptor inhibitor (Active Comparator): Aspirin with P2Y12 receptor inhibitor after 3-month DAPT(aspirin with ticagrelor)
  Interventions: Drug: ticagrelor monotherapy; Drug: Aspirin with P2Y12 receptor inhibitor

INTERVENTIONS:
Drug: ticagrelor monotherapy — • Drug: ticagrelor monothearpy after first 3 months dual therapy
  Other Names: Study group
Drug: Aspirin with P2Y12 receptor inhibitor — • Drug: aspirin plus ticagrelor dual therapy during 12 months
  Other Names: Control group
  Arms: Aspirin with P2Y12 receptor inhibitor

SUMMARY:
To compare the clinical outcomes of dual antiplatelet therapy with aspirin and P2Y12 receptor inhibitor vs. ticagrelor monotherapy at 3 months after PCI in patients with ST-elevation myocardial infarction.

DETAILED DESCRIPTION:
The purpose of this study is to compare the use of ticagrelor alone versus P2Y12 receptor inhibitor and aspirin together after PCI among ST-elevation myocardial infarction patients who complete 3-month course of dual antiplatelet therapy. The object of this study is to determine the effectiveness and safety of ticagrelor alone, compared to P2Y12 receptor inhibitor plus aspirin in reducing clinically relevant bleeding and in reducing ischemic adverse events among patients diagnosed with ST-elevation myocardial infarction undergoing PCI with second-generation drug-eluting stent.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Patients who received new generation sirolimus-eluting (Osiro®) stent implantation for treating ACS
* Provision of informed consent

Exclusion Criteria:

* Age > 80 years
* Pregnant women or women with potential childbearing
* Life expectancy < 1 year

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
NACE: net clinical adverse event | 12 months after randomization
  The sum of major adverse cardiac and cerebrovaascular event(MACCE) and bleeding event(BARC score)
Major adverse cardiac and cerebrovaascular event(MACCE) | 12 months after randomization
  Major adverse cardiac and cerebrovaascular event(MACCE) includes 1)all-cause motality, 2) acute MI, 3)cerebrovascular event, 4)stent thrombosis
Major bleeding (BARC type 3,5) | 12 months after randomization
  The number of participants with first occurrence of clinically relevant bleeding episode, defined as Bleeding Academic Research Consortium (BARC) Types 3 or 5 bleeding. BARC bleeding types range from 0 (no bleeding) to 5 (fatal bleeding).
  type 3a: Overt bleeding plus hemoglobin drop of 3 to < 5 g/dL (provided hemoglobin drop is related to bleed); transfusion with overt bleeding, type 3b: Overt bleeding plus hemoglobin drop < 5 g/dL (provided hemoglobin drop is related to bleed); cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring IV vasoactive agents, type 3c: Intracranial hemorrhage confirmed by autopsy, imaging, or lumbar puncture; intraocular bleed compromising vision, type 5a: Probable fatal bleeding, type 5b: Definite fatal bleeding (overt or autopsy or imaging confirmation in accordance with BARC Definitions

SECONDARY OUTCOMES:
Individual component of MACCE and bleeding episode | 12 months after randomization
  1. All-cause mortality :Individual component of MACCE
  2. Acute MI :Individual component of MACCE
  3. Cerebrovascular event :Individual component of MACCE
  4. Stent thrombosis :Definite or probable stent thrombosis defined by Academic Research Consortium (ARC)
  5. Bleeding :Bleeding Academic Research Consortium (BARC) type 3 or 5

CONTACTS AND LOCATIONS:
Overall Officials: Kyungil Park, Ph.D, Principal Investigator — Dong-A University Hospital
Locations (1):
- Department of Internal Medicine,Dong-A University College of Medicine, Busan, South Korea